CLINICAL TRIAL: NCT00003016
Title: Reliable Assessment of the Efficacy and Safety of Prolonging the Use of Adjuvant Tamoxifen: A Large, Simple, Randomised Study
Brief Title: Prolonged Tamoxifen Compared With Shorter Tamoxifen in Treating Patients Who Have Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Oxford (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000065596; ATLAS; EU-96064
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2002-10

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: tamoxifen citrate
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by reducing the production of estrogen. It is not yet known if prolonged tamoxifen is more effective than shorter tamoxifen therapy following curative treatment for breast cancer.

PURPOSE: This randomized phase III trial is studying giving tamoxifen over a prolonged period of time to see how well it works compared to giving tamoxifen over a shorter period of time in treating patients who have had a breast tumor removed.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the balance of risks and benefits in prolonging the duration of adjuvant tamoxifen by at least 5 years in patients with curatively treated breast cancer who have already had about 5 years of adjuvant tamoxifen.

OUTLINE: This is a randomized study. After about 5 years of adjuvant tamoxifen, recurrence-free patients are randomized to stop tamoxifen treatment immediately or to continue tamoxifen treatment for at least 5 more years.

Patients are followed annually.

PROJECTED ACCRUAL: Approximately 20,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Curatively treated carcinoma of the breast
* Currently taking adjuvant tamoxifen

  * Must be substantial uncertainty as to whether or not to continue tamoxifen (i.e., no clear indication or definite contraindication to further treatment with tamoxifen)

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

Other:

* Not pregnant or nursing
* No contraindications to receiving tamoxifen
* No other serious medical problems

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior biologic therapy allowed

Chemotherapy:

* Prior chemotherapy allowed

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* Prior radiotherapy allowed

Surgery:

* Prior surgery allowed

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20000 (Estimated)
Dates: Start 1995-10

PRIMARY OUTCOMES:
Overall survival (i.e., all-cause mortality)

SECONDARY OUTCOMES:
Specific-cause mortality
Incidence of second primary tumors

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Arriagada, MD, Study Chair — Karolinska Institutet
Locations (1):
- Atlas Trial Office, Oxford, England, United Kingdom